CLINICAL TRIAL: NCT04157374
Title: Action Observation Training in Patients With Chronic Low Back Pain
Acronym: LBP-AOT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patients due to Covid-19 pandemic
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Head of Physiotherapy, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLF19/01
Record Dates: First submitted 2019-08-06; First posted 2019-11-08 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: AOT; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): AOT and Active exercises
  Interventions: Other: Action Observation training; Other: Active Exercises
- Control group (Active Comparator): Active exercises
  Interventions: Other: Active Exercises

INTERVENTIONS:
Other: Action Observation training — They have to watch a video showing a person carrying out exercises (12 exercises: 3 of stretching, 3 of core stability, 3 of mobilization and 3 of functional). then they have to practice them. The observation of the exercises and their performance last 8 minutes (4 minutes for observation and 4 minutes for practice). They have to repeat the exercises 5 times per week for 3 weeks.
  Other Names: AOT
  Arms: EXPERIMENTAL GROUP
Other: Active Exercises — Execution of exercises: 3 of stretching, 3 of core stability, 3 of mobilization and 3 of functional activity. Patients of the control group recieve a brochure with the same exercises the patients of the experimental group received through the video. They will be asked to read the exercise 3 times and to practice it for 4 minutes. They have to repeat the exercises 5 times per week for 3 weeks.

SUMMARY:
The study is a single-blind controlled randomized clinical trial.

DETAILED DESCRIPTION:
Patients will be recruited and then randomly assigned by an external collaborator to the experimental group or to the control group. To the patients that belong to the experimental group will be asked to watch a video showing a person carrying out some exercises (12 exercises: 3 of stretching, 3 of core stability, 3 of mobilization and 3 of functional) and then they will have to practice them.On the other hand, to the patients that belong to the control group will be given a brochure with the same exercises the patients of the experimental group received through the video. Both groups will have to watch the video or read the brochure and repeat the exercises 5 times per week for 3 weeks. Patients will be evaluated before the treatment (T0), three weeks after the beginning (T1) and 4 months upon the end of it (T2). The evaluation will consist in the administration of the Oswestry Disability Index, of the Tampa Scale of Kinesiophobia, of the Numerical Rating Scale and of the Medical Outcomes Study Short Form 36.

A physiotherapist will instruct the patients about the exercises while a second one blinded about the belonging group of patients, will administer the evaluation scales.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic aspecific LBP (documented story of more than 12 week-long symptomatology)
* Good understanding of Italian language
* Aged over 65

Exclusion Criteria:

* Severe sight or hearing impairement
* Cognitive deficit (assessed by a Mini Mental State Examination score ≤21 [14]).
* Specific LBP (previous spine surgery, deformation, infection, fracture, malignant tumor, general disorders or neuromuscular pathologies)
* Patients who previously experimented AOT

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Change of disability of patients | Patients will be evaluated before the treatment (T0), three weeks after the beginning (T1) and 4 months upon the end of it (T2)
  Change in Oswestry Disability Index (ODI-I). Range: 0 (lower disability), 50 (higher disability)

SECONDARY OUTCOMES:
Pain of patients | Patients will be evaluated before the treatment (T0), three weeks after the beginning (T1) and 4 months upon the end of it (T2)
  Numeric rating Scale (NRS), Range: 0 (no pain), 10 (maximum pain)
Quality of life of patients | Patients will be evaluated before the treatment (T0), three weeks after the beginning (T1) and 4 months upon the end of it (T2)
  Short form 36.36 Items divided in 8 sub-scales. Each of the 8 summed scores is linearly transformed onto a scale from 0 (negative health) to 100 (positive health) to provide a score for each subscale. Each subscale is used indipendently.
fear of movement of patients | Patients will be evaluated before the treatment (T0), three weeks after the beginning (T1) and 4 months upon the end of it (T2)
  TAMPA Scale of kinesiophobia, Range: 13 (minimum level of kinesiophobia)- 52 (maximum level of kinesiophobia).

CONTACTS AND LOCATIONS:
Locations (1):
- Roberto Gatti, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT04157374/Prot_SAP_000.pdf